CLINICAL TRIAL: NCT04294342
Title: Health Promotion and Prevention: The Impact of Specifically Adapted Judo-based Training Program on Risk Factors for Falls Among Adults at Work
Brief Title: The Impact of Specifically Adapted Judo-based Training Program on Risk Factors for Falls Among Adults
Acronym: J4BA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalarna University (Other)
Collaborators: Sormland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Michail Tonkonogi, Professor in Medical Science, Dalarna University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: J4B180802-Fallkompetens
Record Dates: First submitted 2020-03-01; First posted 2020-03-04 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Accidental Fall; Fall Injury; Work-related Injury; Work Accident
Keywords: Fall prevention; Physical training; judo; judo4Balance; Break falls; Health and Safety; Falling at work

STUDY DESIGN:
Intervention Model Description: An intervention group which will be training the 10-week judo4 balance
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants in 10 week Judo Inspired Exercise program (Active Comparator): The intervention included 10 sessions, using a 10-week (45-50 minutes /week) pre-established program called Judo4Balance, a structured exercise program which consists of three blocks. All sessions include: Balance, Strength, power and break fall exercises. The intervention group i tested before and after the 10 week exercise.
  Interventions: Behavioral: Active Comparator: Participants in 10 week Judo Inspired Exercise program
- Control Group (No Intervention): The subjects in the control group go about their normal life for 10 weeks without any intervention. The control group is tested before and after the 10 week period.

INTERVENTIONS:
Behavioral: Active Comparator: Participants in 10 week Judo Inspired Exercise program — The intervention included 10 sessions, using a 10-week (45-50 minutes /week) pre-established program called Judo4Balance, a structured exercise program. Each session consisting of warm-up, balance, strength, power and break fall exercises. There is clear a progression within the 10 week program in three main blocks. Block 1: learning the exercises and principle movements, Block 2 more resistance and advance falling techniques, Block 3 Power training and falling strategies from stand up positions.
  Other Names: Judo4Balance: Fall-Preventive Exercise Group
  Arms: Participants in 10 week Judo Inspired Exercise program

SUMMARY:
This is a control study with a 2-group pretest-posttest design investigating the effects of a 10-week judo-inspired exercise program (Judo4Balance) for physical functions, self-efficacy, activity level, and fall techniques among working adults & part-time working retired people.

Falls constitute a common and severe threat to older men and women's health worldwide. However, falls are not just a problem of advanced age, studies have been reporting that falls are a problem at all ages. Nevertheless, falls are under-studied, particularly among young and middle-aged adults (working age adults). For all fall-related injuries among adults, the proportions have been reported to be 32.3% among older adults, 35.3% among middle-aged adults, and 32.3% among younger adults in the United States. This indicates that falls and fall related injuries represent a significant threat to public health at all ages. Therefore, new innovative ways of prevention is much needed and needs to be studied.

DETAILED DESCRIPTION:
The aim of this study is to evaluate and document whether a ten week standardized judo inspired exercise program (Judo4Balance) which include both training the physical qualities such as strength and balance as well as the "break fall" technique can influence the risk of falling as well as reduce the negative consequences of an accidental fall.

Questions asked:

* Can a ten week standardized judo based exercise program improve the "break fall" competence among adults ?
* Can a ten week standardized judo based exercise program improve the fall-efficacy at home and at work among adults ?
* Can a ten week standardized judo based exercise program improve the physical status with regards to the risks for falls among adults ?
* Can a ten week standardized judo based exercise program improve the balance among adults ?
* Could a ten week standardized judo based exercise program be a useful tool in an organisation's preventive Health and Safety work.

The study included two groups with ethical approval to recruit up to 100 individuals in the intervention group and up to 100 individuals in a control group. (control participants are selected mainly the same workplace where the group exercises are being performed and consists of a similar sample of age, sex and physical status ).

The study is conducted in accordance with the Declaration of Helsinki. This study was approved by the Ethical Committee of the Uppsala Region (Dnr 2018/239). Each participant voluntarily provided a written informed consent before participating. Participants were informed that they could withdraw from participation at any time for any reason without any consequences. The participants received no compensation for participating in the study.

A total of seven different workplaces from different parts of Sweden participate in the study of the judo-inspired exercise program (construction and steel industry, healthcare, pre-school, insurance office, advertising, and health and safety consultants). Judo Clubs from different locations in Sweden as well as an insurance company offered the program as part of their preventive Health and Safety at the workplace program. Workplaces report an interest in participating and view their participation as part of their systematic work to promote Health and Safety among employees. Information and an invitation to participate in the 10-week program were provided to employees at the workplace setting.

After an acceptance to participate, written consent is obtained. Measurements were performed at the workplace by a qualified judo instructor.

A total of three qualified Judo instructors, familiar with the physical tests performed the pre- and post-assessments. A total of 14 qualified judo instructors provide instructions in the different groups (on average, 2 instructors per group of 10-18 persons). The instructors teaching the special exercise program are required to have at least a blue belt in judo (which means a minimum of 5 years of regular judo and break fall training). All the instructors teaching the classes in the study have black belts. To teach the program, there are also a requirement to have a coaching license from the Swedish Judo Federation and to have undergone a specific weekend course in the Judo4Balance program, with a focus on teaching judo-related exercises and fall techniques to adult beginners.

The program is delivered in a 45-50-minute session once a week for ten weeks at the respective workplace or other suitable location for the group exercise. The 10 week program is divided into three blocks and taught by experienced and especially trained judo instructors.

Block 1: Good technique during break fall training and strength training, accustomed the body to regular training, find the right level of training for the group, build up load resistance in muscles, tendons and bones. Challenge the balance through new movements not used everyday. Flexibility training for stiff joints such as neck and upper back.

Block 2: Improve "break fall" technique and strength exercises, increase the loads and further challenge the balance and coordination, increase range of motion and introduce "power training".

Block 3: Train the skill of explosive power during strength exercises and break falls. Challenge the balance with increased complexity and difficulty.

The participants both in the intervention group and control group are tested before and after the 10 week period. After the tests have been carried out a questionnaire is to be sent out to the instructors to get their evaluation of the suitability and effectiveness of the program at the work place. A similar questionnaire will be sent out to the participants to evaluate their experience of this preventive program from a Health and Safety at work perspective.

There is strong evidence that exercise can reduce the risk of falling. Nevertheless, judo based training has not to the investigators knowledge been scientifically investigated for working adults with the aim of reducing falls at the workplace and elsewhere. Neither has it been studied if this type of group training is motivational for continuing physical activity after the intervention or for improving the health and safety among employees.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age. Understanding oral and written communication in Swedish.

Exclusion Criteria:

* Physically fragile individuals that are so weak that they cannot sit up without support or not being able to hold up neck when laying on the floor or rolling backwards
* Individuals with aortic aneurysm, angina pectoris or recently has had a cataract operation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in participants "break fall" competence/skill | Before and after 10 weeks of training
  Two tests have been developed to test the skills for falling backwards as well as falling forwards in a safe setting, with progressive difficulty. Four Judo puzzle mats are needed for the test. The "break fall" technique froward and backward are graded from a 0-4 point scale. (where 0 is not being able to lay down and get up from the floor and 4 is being able to fall safely from a standing up position, thus representing the best score).
Change in participants' fall efficacy after 10 weeks | Before and after 10 weeks of training
  The change in falls-efficacy will be measured through - Modified Falls-Efficacy Scale - Falls Efficacy Scale-Swedish version (FES-S) and Falls Efficacy Scale-Swedish version for working age (FES-S-W) is used to measure the self-confidence in the ability to perform various daily activities without falling.The FES-S-W was extended with six additional questions, with the aim to ask people of working age about their confidence related to falling as well as their confidence of not getting hurt when falling. The original instrument consists of 13 items and the extended test 19 items. Each item is rated from 0 to 10, with a maximum score of 130/190 points, which represents the highest level of self-efficacy. The original instrument has been shown to have high test-retest reliability.
Change in Balance | Before and after the 10 weeks of training
  The Mini-BESTest and Mini-BESTest- W were used to measure balance. The original test includes 14 different tasks on 4 subscales. The extended test includes six additional items: feet shoulder-width apart, on toes for extended time (30 seconds); feet together, eyes closed and on toes; walking backwards; walking backwards on a line; standing on one leg on a foam surface left/right; change in gait speed backwards; and step over obstacles backwards. All tasks are graded from 0 to 2 points, with a total maximum score of 28 points for the original test and 40 points for the extended test. The higher the score the better the performance. The original test has high reported test-retest reliability and interrater reliability.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB-W) | Before and after 10 weeks of training
  Short Physical Performance Battery (SPPB) is used to assess the physical performance in the lower extremities, which was expanded with an additional difficulty progression to suit people of working age (W). The additional progression included advanced items in each of the three components: balance (tandem with heel raise, and tandem with heel raise with closed eyes), gait speed (backwards), and lower body power (chair stand on one leg -left/right). The original scale scores range from 0 to 4 for three components, with an additional score of 20 for the additional items. A total score of 12 represents the best performance for the original test and 32 the best score for the expanded test. The original SPPB has shown to predict the risk of falls in adults over the age of 60. The test has shown to have good test-retest reliability and being sensitive to changes.
Change in level of Physical Activity | Before and after 10 weeks training
  Frändin/Grimby Activity Scale is used to measure the level of physical activity. Three different questions are used capturing activity levels during summer, winter, and at the workplace. The scales range from 1 to 6, with 1 representing 'hardly active at all' and 6 representing 'intensive exercise regularly and several times per week.' The original scale has been evaluated and shown to have good validity.
Judo4Balance Instructors perception of the suitability and effectiveness of the program | After the 10 weeks of training
  A questionnaire will be sent out to the instructors to capture their view the exercise program and its effects on the participants and the workplace environment from a workplace practical and Health and Safety perspective. The initial three questions are graded on a scale from 1-10 where 5 represents "meets expecations" and 1 "not at all meet expectations" and 10 " highly exceeds expectations. The last questions are open questions.
Judo4Balance - Participant Survey | After the 10 week program
  An anonymous survey will be sent out to the participants (after training and testing is finished) to catch their perception of the program from a work place "Health and Safety" perspective. Indicators such as: met expectations, team building, continued interest in exercising and joy at the workplace will be asked. The initial questions are graded on a scale from 1-10 where 5 represents "meet expectations or agree" and 1 "not at all meet or agree" and 10 represents "highly exceeds expectations". There are also some open questions.

CONTACTS AND LOCATIONS:
Overall Officials: Michail Tonkonogi, PhD, Principal Investigator — Dalarna University
Locations (1):
- Dalarna University, Falun, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: No
We are currently investigating with regard to the newly introduced GDPR (data integrity) laws within the European Union which individual data that decoded could be possible to share with other researchers and in what format. However, the extended test protocols for adults as well as newly developed test protocols which could have significant impact on improving the research among more physically adept adults with regards to the risk of falls and fall injury could be released for the common good of improving and enhancing the research in this field within 6 months - 1 year after the first publication.

REFERENCES:
- [Result] Timsina LR, Willetts JL, Brennan MJ, Marucci-Wellman H, Lombardi DA, Courtney TK, Verma SK. Circumstances of fall-related injuries by age and gender among community-dwelling adults in the United States. PLoS One. 2017 May 4;12(5):e0176561. doi: 10.1371/journal.pone.0176561. eCollection 2017. PMID 28472065
- [Result] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Result] Franchignoni F, Horak F, Godi M, Nardone A, Giordano A. Using psychometric techniques to improve the Balance Evaluation Systems Test: the mini-BESTest. J Rehabil Med. 2010 Apr;42(4):323-31. doi: 10.2340/16501977-0537. PMID 20461334
- [Result] Hellstrom K, Lindmark B, Wahlberg B, Fugl-Meyer AR. Self-efficacy in relation to impairments and activities of daily living disability in elderly patients with stroke: a prospective investigation. J Rehabil Med. 2003 Sep;35(5):202-7. doi: 10.1080/16501970310000836. PMID 14582550
- [Derived] Arkkukangas M, Baathe KS, Ekholm A, Tonkonogi M. A 10-week judo-based exercise programme improves physical functions such as balance, strength and falling techniques in working age adults. BMC Public Health. 2021 Apr 17;21(1):744. doi: 10.1186/s12889-021-10775-z. PMID 33865349
- See also: Link to the non-profit Swedish Judo Federation Fall Prevention Program — https://judo.se/fallprevention/